CLINICAL TRIAL: NCT07131007
Title: Construction and Evaluation of Tumor Immunotherapy and Organ Damage Early Warning System Based on Multi-omics
Status: Not yet recruiting | Type: Observational
Sponsor: Hebei Medical University Fourth Hospital (Other)
Collaborators: The First Affiliated Hospital of Dalian Medical University (Other); NuoQing Biotechnology (Shanghai) Co., Ltd. (Unknown); Shandong Sanhe Tongyuan Medical Equipment Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024ZD0526105
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-07

CONDITIONS: Malignant Neoplasm; Organ Damage
Keywords: Tumor immunotherapy; Immune checkpoint inhibitors; Immune - related adverse events; organ damage
MeSH Terms: conditions — Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Months
Biospecimen Retention: Samples With DNA — Before medication administration and 7 days after medication administration, blood, urine, and feces of patients will be collected for multi - omics analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tumor Immunotherapy Cohort: Cancer patients receiving immune checkpoint inhibitors (ICIs). We observe their clinical course, collect organ function data, and perform multi - omics analysis to construct an organ damage early - warning system.
  Interventions: Behavioral: Immunotherapy Monitoring and Sample Collection

INTERVENTIONS:
Behavioral: Immunotherapy Monitoring and Sample Collection — For cancer patients receiving immune checkpoint inhibitors (ICIs), we conduct behavioral monitoring: collect blood, urine, and feces samples before medication and 7 days after medication for multi - omics analysis. Monitor organ function indicators at 24 hours, 72 hours, and 1 week post - medication. No interference with standard ICI treatment; focus on observational data collection to construct an organ damage early - warning system.

SUMMARY:
This project is based on the in-depth analysis and integration of multi-omics data, including but not limited to genomics, transcriptomics, proteomics, and metabolomics. It aims to construct a comprehensive early-warning system for organ function damage in immune-related adverse events (irAEs) associated with immune checkpoint inhibitors (ICIs) during tumor immunotherapy. The core objective of this system is to enhance the overall safety and efficacy of tumor immunotherapy.

First, the project leverages a database to mine the differential omics data of tumor immunotherapy patients with combined organ dysfunction (including combined and non-combined severe infections) within the scope of this project. By integrating biochemical indicators and related hemodynamic data, it constructs a risk early-warning system for organ damage in patients undergoing tumor immunotherapy, while verifying its clinical value and guiding significance.

The specific contents mainly include: capturing specific molecules of organ damage in severe patients after tumor immunotherapy, screening genes, proteins, and metabolic products related to organ damage (including the heart, lungs, brain, liver, kidneys, gastrointestinal tract, etc.), and identifying new specific organ damage biomarkers under different pathogenic factors such as tumor immunotherapy, infections, and irAEs. It collects general clinical information, biochemical indicators, and hemodynamic indicators, and combines multi-omics data to establish an organ damage prediction model. Machine learning algorithms are used for optimization to construct an early-warning system.

Model optimization within the system will be carried out, along with prospective clinical research and multi-dimensional verification. By evaluating the accuracy and cost-effectiveness of the model, it provides decision-making support for clinicians and promotes the development of personalized treatment.

ELIGIBILITY:
Inclusion Criteria:

· Patients with cancer who are receiving immune checkpoint inhibitor treatment.

Exclusion Criteria:

* Active phase of severe autoimmune disease.
* Severe organ dysfunction.
* Presence of active infection.
* Pregnancy or lactation.
* Allergy to drug components.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients receiving immune checkpoint inhibitor therapy, excluding those with active autoimmune disease, severe organ dysfunction, or active infection, to evaluate organ damage early - warning signals.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Whether the patient has developed immune-related organ damage and the severity grade of such damage (if it occurs). | 1 month post - organ damage diagnosis
  The severity of immune-related adverse events (irAEs) is graded in accordance with the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, ranging from Grade 1 (mild symptoms) to Grade 5 (death).

SECONDARY OUTCOMES:
Liver injury indicators ：Total Bilirubin (TBIL) | 1 month
Liver injury indicators ：Aspartate Aminotransferase（AST） | 1 month
Liver injury indicators ：Alanine Aminotransferase（ALT） | 1 month
Renal injury indicators： Creatinine (Cr） | 1 month
Renal injury indicators： Neutrophil Gelatinase-Associated Lipocalin (NGAL) | 1 month
Myocardial injury indicators ：High-Sensitivity Troponin T (hs-cTnT) | 1 month
Lung injury indicators ： Krebs von den Lungen-6 (KL-6) | 1 month
Inflammatory indicators： C-Reactive Protein (CRP) | 1 month
Inflammatory indicators：Interleukin-6 (IL-6) | 1 month
Inflammatory indicators： Tumor Necrosis Factor-α (TNF-α) | 1 month
Metabolomics indicators ：hormone levels | 1 month
Metabolomics indicators ：cholesterol | 1 month
Metabolomics indicators ：triglycerides | 1 month
Metabolomics indicators ：blood glucose | 1 month
Multi-omics indicators ： microbiota composition changes | 1 month

IPD SHARING:
Plan to Share IPD: No
To protect the privacy of participants and ensure compliance with ethical guidelines, individual participant data (IPD) contains sensitive information such as medical history and biomarker details. At present, there are no plans to share IPD externally. If future sharing is considered, a formal review process including ethical approval and data de - identification will be implemented.